CLINICAL TRIAL: NCT00594555
Title: A Phase II Study of CLAG Regimen in Combination With Imatinib Mesylate (Gleevec) in Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: A Study Evaluating the Effects of CLAG With Gleevec in Refractory or Relapsed Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator resigned position with the University of Cincinnati, closing study at this site will reopen study in new position
Sponsor: University of Cincinnati (Other)
Collaborators: Novartis (Industry)
Responsible Party: Rami Komrokji, MD, The University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CST1571AU235 / Komrokji; CST1571AUS235
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Myeloid Leukemia, Blast Crisis; Acute Myeloid Leukemia
Keywords: Blood disease, bone marrow; AML; CML,Blast Crisis
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis; Leukemia, Myeloid, Acute; Hematologic Diseases | interventions — Imatinib Mesylate; Cladribine; Cytarabine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm - treatment period (Experimental): Drug Name/Days Administered
  Neupogen/Days 1-6
  CLAG/Days 2-6
  Gleevec/Days 2-15
  Interventions: Drug: Imatinib Mesylate; Drug: CLAG

INTERVENTIONS:
Drug: Imatinib Mesylate — Imatinib Mesylate: 400mg po BID every day. Imatinib Mesylate will be administered Day 2 to Day 15
  Other Names: Gleevec (Imatinib Mesylate)
Drug: CLAG — Cladribine: 5mg/m2 administered through a 2 hour intravenous infusion daily for 5 consecutive days starting on Day 2
  Cytarabine: 2gm/m2 administered through a 4 hour intravenous infusion starting 2 hours after the ignition of Cladribine for 5 days starting on Day 2
  G-CSF: 300mcg sc for 6 days starting at 24 hours (Day 1) before the first dose of Cladribine; administration starting on Day 1 for 6 days
  Other Names: Cladribine, Cytarabine & G-CSF (also know as CLAG)

SUMMARY:
The purpose of this study is to evaluate the safety of combined chemotherapy treatment (CLAG regimen) with Imatinib Mesylate (Gleevec) in patients with AML.

DETAILED DESCRIPTION:
In relapsed or resistant acute myeloid leukemia (type of blood cancer where immature blood cells are increased, blocking normal blood cells production) no standard therapy exits. Response rates are similar for different chemotherapy treatments. Allogenic stem cell transplant remains the only curative option

The purpose of this study is to evaluate the safety of combined chemotherapy treatment (CLAG regimen) with Imatinib Mesylate (Gleevec). The CLAG regimen is a combination of the chemotherapy drugs cladribine and cytarabine, as well as, neupogen which increases the white blood counts.

Imatinib Mesylate is believed to work by interfering with the abnormal protein by blocking it from telling the body to keep making more and more abnormal white blood cells. Imatinib Mesylate is approved by the FDA for the treatment of chronic myeloid leukemia (CML) and some types of acute lymphoblastic leukemia (ALL). Its use in combination with CLAG regimen is considered experimental for the treatment of Acute Myeloid Leukemia / CML blast crisis

The goal of the study is to find out what effects (good and bad) Imatinib Mesylate (Gleevec)combined with chemotherapy (CLAG regimen) on acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria

* Men and Women of all ethnic groups whose age is ≥ 18 years old.
* Diagnosis of AML or CML blast crisis, according to WHO criteria, except acute promyelocytic leukemia AML-M3 FAB subgroup.
* Refractory or Relapsed AML.

  * Refractory AML is defined as failure to achieve CR after 2 cycles of induction chemotherapy or persistent (>40%) bone marrow blasts after one cycle of chemotherapy induction.
  * Relapsed AML is defined as any evidence of disease recurrence after achieving CR. Early relapse is defined as that occurring within 12 months and late relapse is defines as that occurring after 12 months.
* ECOG performance status of 0 or 1.
* Patients must sign a written informed consent.
* Females of childbearing potential must not be pregnant or actively nursing a child. They must have a negative pregnancy test 7 days before initiation of study drug administration.
* Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Male and females of reproductive potential must agree to employ an effective barrier method of birth control throughout the duration of the trial and for 3 months following study medication discontinuation.

Exclusion Criteria

* Abnormal Kidney Functions: creatinine ≥2.5mg/dL; if creatinine is between 2.0-2.5, patient should have GFR measured and the dose of Cytarabine may be adjusted accordingly.
* Abnormal Liver Functions: Bilirubin .2mg/dL, transaminases (AST/ALT) more that 2.5 times the institutional upper limits of normal (IULN)
* Systemic active infection, unless controlled on active therapy.
* Patients with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria ( i.e., congestive heart failure, myocardial infarction within 6 months of the study), EF 30%.
* Patient has known chronic liver disease (i.e., chronic active hepatitis and cirrhosis).
* Patient has known diagnosis of human immunodeficiency virus (HIV) infection.
* History of other curatively untreated malignancy, except non-melanotic skin cancers.
* Patients that have received investigational agents within 1 month of study entry.
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to Gleevec or any component of the CLAG regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Establishing the overall response rate and the safety of combining imatinib mesylate with CLAG regimen | The amount of time it takes to enroll 20 pts. About 1 year

SECONDARY OUTCOMES:
The sample size is calculated based on two stage Phase II clinical design. Ten patients will be accrued during stage 1 and 10 during stage 2). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rami S Komrokji, MD, Principal Investigator — The University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States